CLINICAL TRIAL: NCT00477373
Title: Gulf Evaluation of VAlproate (Depakine Chrono) in maNia Study
Acronym: GEVANS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DPKOT_L_01567
Record Dates: First submitted 2007-05-22; First posted 2007-05-23 (Estimated); Last update posted 2008-12-19 (Estimated); Status verified 2008-12

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): If the daily dose does not exceed 1000 mg, Depakine CHRONO can be administered once a day. If the dose is greater than 1000 mg/day, Depakine CHRONO will be administered in a bid regimen: one tablet in the morning and one tablet in the evening.
  Interventions: Drug: depakine chrono

INTERVENTIONS:
Drug: depakine chrono — Depakine Chrono 500 mg

SUMMARY:
To assess the efficacy of Di-valproate in Bipolar I patients suffering from a manic episode according to DSM IV (APA 1994) over a 12 weeks period of treatment.

To evaluate the clinical safety of Di-valproate.

ELIGIBILITY:
Inclusion Criteria:

* In or out patients
* Patients with a current diagnosis of Bipolar I Disorder according to DSM IV (296)
* Patients suffering from a current manic episode or mixed episode

Exclusion Criteria:

* Patients who participated in a clinical trial within the three preceding months
* Patients with a history of valproate intolerance defined as valproate discontinuation due to medically significant adverse effects.
* Patients with a CNS neoplasm, demyelinating disease, degenerative neurological disorder, active CNS infection or any progressive disorder
* Patients with a history of seizure disorder, cerebral vascular disease, structural brain damage from trauma, clinically significant focal neurological abnormalities, known EEG with frank paroxysmal activity or a known CT scan of the brain demonstrating gross structural abnormalities
* Patients with uncontrolled gastro-intestinal, renal, hepatic, endocrine, cardiovascular, pulmonary, immunological or hematological disease
* Patients with acute or chronic hepatitis
* Patients with current or past pancreatitis
* Patients with recent history (3 months or less) of substance or alcohol dependence according to DSM IV
* Pregnancy or lactation. Women of child bearing age should be using a reliable contraceptive method
* Patients that require more than 325 mg of aspirin per day
* Patients with a medical condition which requires the continuous use of medication which could interfere with the evaluation of safety or efficacy of valproate : anticonvulsant or anticoagulant therapy, MAO inhibitors, zidovudine
* Patients having received any depot neuroleptic within six weeks prior to baseline
* Patients who received antidepressant drugs within 5 days before baseline and patients who received fluoxetine within 20 days
* Patients judged by the investigator to have serious risk of suicide
* Patients necessitating an Electro Convulsive Therapy

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2006-12; Primary Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The mean change in the Clinical Global Impressions Scale for Bipolar Disorder (CGI-BP)Severity score as well as the change in CGI-BP. | D0, D21 and D-end

SECONDARY OUTCOMES:
Percentage of responders defined by a decrease of at least 50% of the CGI-BP. | D0 and D-end
Percentage of responders defined by a decrease of at least 50% of the CGI-BP. | D0 and D21
Time to achieve 50% and 30% improvement in the CGI-BP score. | From randomization to the end of the study
Time to a sustained improvement in the CGI-BP. | From randomization to the end of the study
Time to antidepressants use. | From randomization to the end of the study
Time to drop-out for any reason. | From randomization to the end of the study
Safety :Occurrence of any side effect leading to treatment discontinuation. | From inform consent signed until patient's recovery or stabilization

CONTACTS AND LOCATIONS:
Overall Officials: Hisham - MAHMOUD, MD, Study Director — Sanofi-aventis administrative office Gulf
Locations (4):
- Sanofi-aventis administrative office, Bahrain, Bahrain
- Sanofi-aventis administrative office, Kuwait City, Kuwait
- Sanofi-Aventis Administrative Office, Muscat, Oman
- Sanofi-aventis administrative office, Qatar, Qatar